CLINICAL TRIAL: NCT03269955
Title: The Effect of Application of Fibrinogen/Thrombin-coated Collagen Patch (TachoSil®) in Pancreaticojejunostomy for Prevention of Pancreatic Fistula After Pancreatoduodenectomy
Brief Title: The Effect of Application of TachoSil® in Pancreatoduodenectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jae Hoon Lee, M.D, Ph.D, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-0791
Record Dates: First submitted 2017-08-23; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Neoplasm; Pancreatic Periampullary Cancer; Pancreatic Bordeline Tumor
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fibrinogen; TachoSil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- application of TachoSil® (Experimental): Fibrinogen/thrombin-coated collagen patch (TachoSil®) and fibrin glue are applied to the pancreas anastomosis site in pancreatoduodenectomy
  Interventions: Drug: Fibrinogen/thrombin-coated collagen patch
- control (No Intervention): Only fibrin glue alone is applied to the pancreas anastomosis site in pancreaticoduodenectomy.

INTERVENTIONS:
Drug: Fibrinogen/thrombin-coated collagen patch — Tachosil® is cut in half and applied to the front and back of the pancreaticojejunostomy respectively, and fibrin glue is applied on it
  Other Names: TachoSil®
  Arms: application of TachoSil®

SUMMARY:
Fibrinogen/thrombin-coated collagen patch (TachoSil®) is known to have the effect of strengthening tissue anastomosis and promoting suturing to prevent leakage. The purpose of this study is to compare the incidence of pancreatic fistula that is most crucial for surgical outcome and complications in pancreaticoduodenectomy with those of the control group and the TachoSil® apply group.

Patients who were planned to undergo pancreaticoduodenectomy without a history of chronic pancreatitis are enrolled in this open-label, single-center, randomized, single-blind, phase 4 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance score of 0-2
* Periampulary cancer or borderline tumor that is able to resection on preoperative examination
* Patients without distance metastasis
* Bone marrow function: WBC at least 3,000/mm3 or absolute neutrophil count at least 1,500/mm3, Platelet count at least 125,000/mm3
* Liver function: AST/ALT less than 3 times upper limit of normal
* Kidney function: Creatinine no greater than 1.5 times upper limit of normal
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with distant metastases are not eligible
* Recurred periampulary cancer
* Pregnant and breastfeeding women
* Patients with active or uncontrolled infection
* Patients with uncontrolled heart disease
* Patients with moderate or severe comorbidities who are thought to have an impact on quality of life or nutritional status (Liver cirrhosis, chronic kidney failure, heart failure, etc.)
* Patients who underwent other major abdominal organs surgery except for scheduled pancreatoduodenectomy (gastrectomy, colonic resection, etc.)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of pancreatic fistula | At 3 days after surgery
  The evaluation of the pancreatic fistula was based on the international study group of pancreatic fistula (ISGPF). According to the criteria, evaluation of pancreatic fistula was evaluated by measuring the amylase level of the drain tube on the third postoperative day, and the pancreatic fistula was judged to be present when the amylase level was three times higher than the normal level of the amylase in the blood.
Incidence of clinically relevant pancreatic fistula | At 5 days after surgery
  The grade uses ISGPF grading, while the grades B and C are clinically relevant pancreatic fistula. All patients underwent abdominal CT at 5 days postoperatively for grade evaluation.

SECONDARY OUTCOMES:
Incidence of complication except for pancreatic fistula | Through study completion, an average of 1 year
  Complications other than pancreatitis include all complications after pancreatoduodenectomy. Delayed gastric emptying and postoperative bleeding complied with the criteria of the International Study Group, and the severity of complications is classified through the Clavien-Dindo classification.
Removal time of drainage | From date of surgery until the date of the last drainage removal, whichever came first, assessed up to study completion, an average of 1 year
  The timing of removal of the drain tube is determined based on the time of removal of the last drain tube. The removal of the drain tube is assessed at the discretion of the surgeon.
Death | From date of surgery to 30 days after discharge
  The results are for patients who died during hospitalization. If a patient is discharged within 30 days of discharge, the death rate is the same as during death.
Re-admission rate | Through study completion, an average of 1 year
  Includes all cases of re-admission after discharge due to problems associated with pancreatoduodenectomy. Except for cases not related to pancreaticoduodenectomy.
Period of hospitalization after surgery | From date of surgery until the date of discharge, whichever came first, assessed up to study completion, an average of 1 year
  The duration of the hospital stay is calculated based on the time when the actual patient is discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Jaehoon Lee, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpagu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Suzuki Y, Fujino Y, Ajiki T, Ueda T, Sakai T, Tanioka Y, Kuroda Y. No mortality among 100 consecutive pancreaticoduodenectomies in a middle-volume center. World J Surg. 2005 Nov;29(11):1409-14. doi: 10.1007/s00268-005-0152-4. PMID 16222456
- [Background] Bassi C, Butturini G, Molinari E, Mascetta G, Salvia R, Falconi M, Gumbs A, Pederzoli P. Pancreatic fistula rate after pancreatic resection. The importance of definitions. Dig Surg. 2004;21(1):54-9. doi: 10.1159/000075943. Epub 2003 Dec 30. PMID 14707394
- [Background] Benzoni E, Zompicchiatti A, Saccomano E, Lorenzin D, Baccarani U, Adani G, Noce L, Uzzau A, Cedolini C, Bresadola F, Intini S. Postoperative complications linked to pancreaticoduodenectomy. An analysis of pancreatic stump management. J Gastrointestin Liver Dis. 2008 Mar;17(1):43-7. doi: 10.1007/s11749-008-0106-x. PMID 18392243
- [Background] de Castro SM, Kuhlmann KF, Busch OR, van Delden OM, Lameris JS, van Gulik TM, Obertop H, Gouma DJ. Incidence and management of biliary leakage after hepaticojejunostomy. J Gastrointest Surg. 2005 Nov;9(8):1163-71; discussion 1171-3. doi: 10.1016/j.gassur.2005.08.010. PMID 16269388
- [Background] Bassi C, Falconi M, Molinari E, Mantovani W, Butturini G, Gumbs AA, Salvia R, Pederzoli P. Duct-to-mucosa versus end-to-side pancreaticojejunostomy reconstruction after pancreaticoduodenectomy: results of a prospective randomized trial. Surgery. 2003 Nov;134(5):766-71. doi: 10.1016/s0039-6060(03)00345-3. PMID 14639354
- [Background] Govindarajan A, Tan JC, Baxter NN, Coburn NG, Law CH. Variations in surgical treatment and outcomes of patients with pancreatic cancer: a population-based study. Ann Surg Oncol. 2008 Jan;15(1):175-85. doi: 10.1245/s10434-007-9601-7. Epub 2007 Oct 2. PMID 17909913
- [Background] Satoi S, Toyokawa H, Yanagimoto H, Yamamoto T, Yamao J, Kim S, Matsui Y, Takai S, Mergental H, Kamiyama Y; Department of Surgery, Kansai Medical University, Osaka, Japan. A new guideline to reduce postoperative morbidity after pancreaticoduodenectomy. Pancreas. 2008 Aug;37(2):128-33. doi: 10.1097/MPA.0b013e318162cb53. PMID 18665071
- [Background] Peng SY, Wang JW, Lau WY, Cai XJ, Mou YP, Liu YB, Li JT. Conventional versus binding pancreaticojejunostomy after pancreaticoduodenectomy: a prospective randomized trial. Ann Surg. 2007 May;245(5):692-8. doi: 10.1097/01.sla.0000255588.50964.5d. PMID 17457161
- [Background] Fernandez-Cruz L, Belli A, Acosta M, Chavarria EJ, Adelsdorfer W, Lopez-Boado MA, Ferrer J. Which is the best technique for pancreaticoenteric reconstruction after pancreaticoduodenectomy? A critical analysis. Surg Today. 2011 Jun;41(6):761-6. doi: 10.1007/s00595-011-4515-1. Epub 2011 May 28. PMID 21626319
- [Background] Shrikhande SV, Barreto G, Shukla PJ. Pancreatic fistula after pancreaticoduodenectomy: the impact of a standardized technique of pancreaticojejunostomy. Langenbecks Arch Surg. 2008 Jan;393(1):87-91. doi: 10.1007/s00423-007-0221-2. Epub 2007 Aug 17. PMID 17703319
- [Background] Mita K, Ito H, Fukumoto M, Murabayashi R, Koizumi K, Hayashi T, Kikuchi H, Kagaya T. A fibrin adhesive sealing method for the prevention of pancreatic fistula following distal pancreatectomy. Hepatogastroenterology. 2011 Mar-Apr;58(106):604-8. PMID 21661439
- [Background] Chirletti P, Caronna R, Fanello G, Schiratti M, Stagnitti F, Peparini N, Benedetti M, Martino G. Pancreaticojejunostomy with application of fibrinogen/thrombin-coated collagen patch (TachoSil) in Roux-en-Y reconstruction after pancreaticoduodenectomy. J Gastrointest Surg. 2009 Jul;13(7):1396-8; author reply 1399-400. doi: 10.1007/s11605-009-0894-7. Epub 2009 Apr 18. No abstract available. PMID 19381733
- [Background] Simo KA, Hanna EM, Imagawa DK, Iannitti DA. Hemostatic Agents in Hepatobiliary and Pancreas Surgery: A Review of the Literature and Critical Evaluation of a Novel Carrier-Bound Fibrin Sealant (TachoSil). ISRN Surg. 2012;2012:729086. doi: 10.5402/2012/729086. Epub 2012 Sep 13. PMID 23029624
- [Background] Montorsi M, Zerbi A, Bassi C, Capussotti L, Coppola R, Sacchi M; Italian Tachosil Study Group. Efficacy of an absorbable fibrin sealant patch (TachoSil) after distal pancreatectomy: a multicenter, randomized, controlled trial. Ann Surg. 2012 Nov;256(5):853-9; discussion 859-60. doi: 10.1097/SLA.0b013e318272dec0. PMID 23095631
- [Background] Pavlik Marangos I, Rosok BI, Kazaryan AM, Rosseland AR, Edwin B. Effect of TachoSil patch in prevention of postoperative pancreatic fistula. J Gastrointest Surg. 2011 Sep;15(9):1625-9. doi: 10.1007/s11605-011-1584-9. Epub 2011 Jun 14. PMID 21671113
- [Derived] Kwon J, Shin SH, Lee S, Park G, Park Y, Lee SJ, Lee W, Song KB, Hwang DW, Kim SC, Lee JH. The Effect of Fibrinogen/Thrombin-Coated Collagen Patch (TachoSil(R)) Application in Pancreaticojejunostomy for Prevention of Pancreatic Fistula After Pancreaticoduodenectomy: A Randomized Clinical Trial. World J Surg. 2019 Dec;43(12):3128-3137. doi: 10.1007/s00268-019-05172-y. PMID 31502003